CLINICAL TRIAL: NCT02725996
Title: By Using Adoptive Transfer of Autologous NK Cells to Prevent Recurrence of Hepatocellular Carcinoma After Curative Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Zhi Yang, Researcher of Biotherapy Center, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMMU-BTC-006
Record Dates: First submitted 2016-03-28; First posted 2016-04-01 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Natural Killer cells
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- curative therapy+NK infusion (Experimental): Adjuvant adoptive immune therapy using NK cell 4 times after curative therapy
  Interventions: Biological: NK cells; Other: Curative therapy
- curative therapy (Other): Patients who had undergone curative treatment(surgical resection or radiofrequency ablation[RFA]) for HCC of pretreatment clinical stage I or II according to the American Joint Committee on Cancer staging system(6th edition) based on radiologic imaging studies were eligible for this study with no adjuvant treatment
  Interventions: Other: Curative therapy

INTERVENTIONS:
Biological: NK cells — Adjuvant adoptive immune therapy using NK cell 4 times
  Other Names: natural killer cell infusion
  Arms: curative therapy+NK infusion
Other: Curative therapy — Patients who had undergone curative treatment(surgical resection or radiofrequency ablation for HCC of pretreatment clinical stage I or II were eligible for this study with no adjuvant treatment

SUMMARY:
To prove that the efficacy and safety of 'NK group' is superior to 'non-treatment group(Control group)' in patient undergone curative resection(RFA or operation) for hepatocellular carcinoma in China.

DETAILED DESCRIPTION:
No adjuvant therapy has been shown to extend the survival of patients with hepatocellular carcinoma receiving curative treatment.We investigated whether injections of NK cells prolongs recurrence-free survival of patients after curative therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Prior to the test, patient is fully explained about the purpose/ contents and characteristics of the testing medication, and the patient him(her)self, the guardian or the legal representative signed on written consent.
2. Gender unlimited, age from 18 years to 70 years
3. The patient is diagnosed as hepatocellular carcinoma by pathological/ radiological test and he (she) is in the stage of I or II. (refer to the attached file 10). Hepatocellular carcinoma should be shown by radiological test; on dynamic CT, dynamic MRI or on angiography.
4. Child-Pugh Score should be less than 6
5. No matter how the patient has been treated before, his (her) tumor should be totally removed by curative resection (RFA or operation). (based on the agreement date for written consent)
6. Patients must have adequate cardiac function(no cardiac disease, LVEF≥40% ), adequate pulmonary function as indicated by room air oxygen saturation of >94%, and adequate renal function(Cr≤133umol/L).
7. Patient's remaining life-time should be expected at least more than 3 months.

Exclusion Criteria:

1. Hepatocellular carcinoma has been transferred by pathological/ radiological test (Stage III or Stage IV, refer to the exhibit 10)
2. The carcinoma has been invaded to main portal vein or major branch hepatic vein
3. Child-Pugh score is over 6
4. Patient has serious problem with pulmonary function by sub- investigator's opinion
5. Patient who has disease history of immune deficiency
6. Diagnosed as an immune deficiency patient
7. Patient who has disease history of malignant tumor within 5 years before this clinical trial.
8. Patient who had anti-cancer medication before the clinical trial
9. Patient has serious allergic-history by sub- investigator's opinion
10. Patient has serious mental disease by sub- investigator's opinion
11. Pregnant women, nursing mother or having intention of being pregnant during the clinical test
12. Patient who participated in other clinical trial within 4 weeks before this clinical trial
13. Patient who is incongruent to this clinical trial by sub- investigator's opinion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Recurrence Free Survival(RFS) :RFS was measured from the date of randomization to the first recurrence or to death from any cause. | 3 years
Overall Survival(OS) :Overall survival was measured from the date of randomization until death from any cause. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Qian, MD, PhD, Study Chair — Biotherapy Center of Southwest Hospital
Locations (1):
- Southwest Hospital of Third Millitary Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided